CLINICAL TRIAL: NCT05686772
Title: A Better Understanding of the Association Between Problem Gambling and Psychotic Disorders in Young Adults: a New Path Towards Recovery
Brief Title: Prospective Multicenter Cohort Study Evaluating the Incidence and Risk Factors for Problem Gambling Among Young Adults With First-episode Psychosis
Acronym: ANTE-UP
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Olivier Corbeil, PharmD, MSc, Pharmacist, Principal Investigator, Laval University
Other Study IDs: 2020-OJUR-286304
Record Dates: First submitted 2022-12-29; First posted 2023-01-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Gambling Disorder; Psychotic Disorders
Keywords: Gambling; Psychotic disorder; Schizophrenia; Cohort; Multicenter; Prospective; Observational; Incidence; Risk factors
MeSH Terms: conditions — Gambling; Psychotic Disorders; Schizophrenia | interventions — Social Class

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- First-episode psychosis patients: All patients aged 18-35 years with a diagnosis of FEP admitted at two FEP programs in the province of Quebec, Canada.
  Interventions: Drug: Antipsychotic use; Other: Psychiatric comorbidities; Other: Sociodemographics/socioeconomic status; Other: Gambling history; Other: Clinical variables

INTERVENTIONS:
Drug: Antipsychotic use — Use of first/second generation antipsychotics, use of third-generation antipsychotics, use of aripiprazole specifically
Other: Psychiatric comorbidities — Substance use disorders, cluster B personality disorders, anxiety disorder, major depressive disorder, attention-deficit/hyperactivity disorder, tobacco smoking
Other: Sociodemographics/socioeconomic status — Age, gender identity, ethnicity, highest educational attainment, employment, at school, homelessness, in a relationship
Other: Gambling history — Non-problematic gambling at the time of admission and/or previous 12 months
Other: Clinical variables — Main psychiatric diagnosis, history of psychiatric hospitalizations, severity of illness (CGI-S), functioning (SOFAS), concomitant psychotropic medications use

SUMMARY:
The aims of this propsective cohort study are to get a better understanding of the association between problem gambling and psychotic disorders among young adults with first-episode psychosis.

The main questions to be answered are:

1. What is the incidence of problem gambling in this population?
2. What are the predictors of problem gambling in this population?

To do so, putative predictors of problem gambling will be analyzed using Cox regression models:

* Sociodemographics (e.g., age, gender identity, ethnicity, level of education, employment);
* Psychiatric comorbidities (e.g., substance use disorders, cluster B personality disorders);
* Antipsychotic use (first/second-generation, third-generation [aripiprazole, brexpiprazole, cariprazine]);
* Prior gambling history.

DETAILED DESCRIPTION:
All Cox regression models will be adjusted for site-effect. Further multivariable models will be constructed to examine the association between antipsychotic use (as continuous exposure) and incident PBG using the directed acyclic graphs approach to adjust for confounders.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old;
* Diagnosis of first-episode psychosis (i.e., DSM-5 diagnosis of schizophrenia spectrum and other psychotic disorders, as well as DSM-5 bipolar disorder with psychotic features).

Exclusion Criteria:

* Active/prior PBG at te time of admission;
* Loss to follow-up within first three months;
* DSM-5 diagnosis of psychotic disorder due to a medical condition;
* Severe intellectual disability.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients meeting the inclusion/exclusion criteria admitted to 2 first-episode psychosis programs located in Quebec (Canada) during the study period (i.e., November 1st, 2019 - May 1st, 2023).
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Problem gambling | Outcome assessed at every 6-month time point, from patients admission until the first occurrence of the primary outcome, loss to follow-up, or May 1, 2023.
  i) Diagnosis of gambling disorder according to DSM-5 criteria, established by the treating psychiatrist, and/or; ii) Problem gambling according to a score of 8 and more on the Problem Gambling Severity Index, as questioned by the clinical case manager and/or treating psychiatrist

OTHER OUTCOMES:
Sensitivity analysis restricted to DSM-5 gambling disorder | Outcome assessed at every 6-month time point, from patients admission until the first occurrence of the primary outcome, loss to follow-up, or May 1, 2023.
  DSM-5 diagnosis of gambling disorder by treating psychiatrist

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal University Hospital Center, Montreal, Quebec
  - Quebec Mental Health University Institute, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
The participants of this study did not give written consent for their data to be shared publicly, so due to the sensitive nature of the research supporting data is not available.

REFERENCES:
- [Background] Corbeil O, Corbeil S, Dorval M, Carmichael PH, Giroux I, Jacques C, Demers MF, Roy MA. Problem Gambling Associated with Aripiprazole: A Nested Case-Control Study in a First-Episode Psychosis Program. CNS Drugs. 2021 Apr;35(4):461-468. doi: 10.1007/s40263-021-00801-4. Epub 2021 Mar 13. PMID 33713298
- [Background] Corbeil O, Corbeil S, Giroux I, Jacques C, Dorval M, Demers MF, Roy MA. Problem Gambling Associated With Aripiprazole in First-Episode Psychosis Patients: A Series of 6 Case Reports. J Clin Psychopharmacol. 2020 Mar/Apr;40(2):191-194. doi: 10.1097/JCP.0000000000001177. PMID 32134855
- [Background] Lachance A, Corbeil O, Corbeil S, Chalifour G, Breault AS, Roy MA, Demers MF. Case Reports of Aripiprazole and Problematic Gambling in Schizophrenia: A Critical Review of the Evidence. J Clin Psychopharmacol. 2019 Jul/Aug;39(4):393-397. doi: 10.1097/JCP.0000000000001068. PMID 31206391
- [Background] Desai RA, Potenza MN. A cross-sectional study of problem and pathological gambling in patients with schizophrenia/schizoaffective disorder. J Clin Psychiatry. 2009 Sep;70(9):1250-7. doi: 10.4088/JCP.08m04359. Epub 2009 Jun 16. PMID 19538900
- [Background] Haydock M, Cowlishaw S, Harvey C, Castle D. Prevalence and correlates of problem gambling in people with psychotic disorders. Compr Psychiatry. 2015 Apr;58:122-9. doi: 10.1016/j.comppsych.2015.01.003. Epub 2015 Jan 15. PMID 25684263
- [Background] Bergamini A, Turrina C, Bettini F, Toccagni A, Valsecchi P, Sacchetti E, Vita A. At-risk gambling in patients with severe mental illness: Prevalence and associated features. J Behav Addict. 2018 Jun 1;7(2):348-354. doi: 10.1556/2006.7.2018.47. Epub 2018 Jun 5. PMID 29865864
- [Derived] Corbeil O, Soulard M, Huot-Lavoie M, Bechard L, Fournier E, Brodeur S, Essiambre AM, Desmeules C, Theriault C, Abdel-Baki A, Jacques C, Giroux I, Dorval M, Roy MA, Demers MF. Problem gambling among people with first-episode psychosis: protocol for a prospective multicenter cohort study. BMC Psychiatry. 2023 Apr 25;23(1):287. doi: 10.1186/s12888-023-04741-9. PMID 37098506